CLINICAL TRIAL: NCT05166161
Title: A Phase 3 Open-Label Study of PTC923 (Sepiapterin) in Phenylketonuria
Brief Title: A Long-Term Safety Study of PTC923 in Participants With Phenylketonuria
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC923-MD-004-PKU; 2021-000497-28 (EudraCT Number); 2023-509229-31-00 (Other: CTIS Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — sepiapterin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTC923 (Experimental): Participants will receive PTC923 7.5 mg/kg (participants 0 to <6 months of age), 15 mg/kg (participants 6 to <12 months of age), 30 mg/kg (participants 12 months to <2 years of age), or 60 mg/kg (participants ≥2 years of age) orally once daily for a minimum of 12 months or until participant experiences lack of efficacy, adverse events (AEs) that lead to discontinuation, withdraws from treatment, or PTC923 is authorized and commercially available in the specific country.
  Interventions: Drug: PTC923

INTERVENTIONS:
Drug: PTC923 — PTC923 powder for oral use will be suspended in water or apple juice prior to administration.
  Other Names: Sepiapterin; Sephience

SUMMARY:
The main purpose of this study is to evaluate the long-term safety of PTC923 in participants with phenylketonuria, and to evaluate the changes from baseline in dietary phenylalanine (Phe)/protein consumption.

DETAILED DESCRIPTION:
Eligible participants are:

Feeder participants: those who have completed a Phase 3 PTC Therapeutics (PTC) sponsored feeder study.

Non-feeder controlled participants: those who have not completed a feeder study and have blood Phe levels <360 μmol/L at study entry.

Non-feeder uncontrolled participants: those who have not completed a feeder study and have blood Phe levels ≥360 μmol/L at study entry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PKU with hyperphenylalaninemia (HPA) documented by past medical history of at least 2 blood Phe measurements ≥600 μmol/L.
* Women of childbearing potential must have a negative pregnancy test at screening and agree to abstinence or the use of at least one highly effective form of contraception for the duration of the study, and for up to 90 days after the last dose of the study drug.
* Males who are sexually active with women of childbearing potential who have not had a vasectomy must agree to use a barrier method of birth control during the study and for up to 90 days after the last dose of study drug. Males must also refrain from sperm donations during this time period.
* Willing to continue current diet unchanged while participating in the study (unless specifically instructed to change diet during the study by the investigator).

Exclusion Criteria:

* Inability to tolerate oral medication.
* A female who is pregnant or breastfeeding, or considering pregnancy.
* Serious neuropsychiatric illness (for example, major depression) not currently under medical control, that in the opinion of the investigator or PTC, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant.
* Past medical history and/or evidence of renal impairment and/or condition including moderate/severe renal insufficiency (glomerular filtration rate [GFR] <60 milliliters [mL]/minute [min] min as estimated most recently during qualifying participation in a feeder study) and/or under care of a nephrologist.
* Any other condition that in the opinion of the investigator or PTC, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant.
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (for example, methotrexate).
* Concomitant treatment with tetrahydrobiopterin (BH4) supplementation (for example, sapropterin dihydrochloride, KUVAN) or pegvaliase-pqpz (PALYNZIQ).

Additional criteria for non-feeder participants who did not participate in a feeder study:

* Gastrointestinal disease (such as irritable bowel syndrome, inflammatory bowel disease, chronic gastritis, and peptic ulcer disease, etc) that could affect the absorption of study drug.
* History of gastric surgery, including Roux-en-Y gastric bypass surgery or an antrectomy with vagotomy, or gastrectomy.
* History of allergies or adverse reactions to synthetic BH4 or sepiapterin.
* Any clinically significant laboratory abnormality as determined by the investigator.
* Any abnormal physical examination and/or laboratory findings indicative of signs or symptoms of renal disease, including calculated GFR <60 milliliters (mL)/minute/1.73 square meter (m^2).

Confirmed diagnosis of a primary BH4 deficiency as evidenced by biallelic pathogenic mutations in 6-pyruvoyltetrahydropterin synthase, recessive GTP cyclohydrolase I, sepiapterin reductase, quinoid dihydropteridine reductase, or pterin-4-alphacarbinolamine dehydratase genes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (TEAEs) | Baseline up to end of study (up to 4 years)
  A TEAE is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease in a study participant who is administered study drug in this study
Change From Baseline in Dietary Phe/Protein Consumption at Week 26, Measured During Phe Tolerance Assessment Period | Baseline, Week 26
  Phe tolerance is defined as the total amount of dietary Phe (milligrams [mg]/kilogram [kg] per day) ingested while maintaining blood Phe levels within the range of 40 to 360 micromoles (μmol)/liter (L) (defined as ≥40 to <360 μmol/L).

SECONDARY OUTCOMES:
Change From Baseline in Quality of Life (QOL) Using Phenylketonuria-Quality of Life (PKU-QOL) Questionnaire at Months 8, 14, 20, 26, 32, and 38 | Baseline, Months 8, 14, 20, 26, 32, and 38
  QOL using PKU-QOL questionnaire will be assessed in the subset of participants who are able to complete the PKU-QOL (that is, participants whose primary language is English [British or American], Turkish, Dutch, German, Spanish, Italian, Portuguese, or French) (ages 6 to 8 years Parent PKU-QOL; ages 9 to 11 years Child PKU-QOL; ages 12 to 17 years Adolescent PKU-QOL; ages ≥18 years Adult PKU-QOL).
Change From Baseline in QOL Using the European Quality of Life - 5 Dimensions (EQ-5D) at Months 8, 14, 20, 26, 32, and 38 | Baseline, Months 8, 14, 20, 26, 32, and 38
  QOL will be assessed using the EQ-5D (EQ-5D-Y Proxy Version 1 [3 to 7 years]; EQ-5D-Y [8 to 15 years]; EQ-5D-5L ([≥16 years]).
Palatability of PTC923 | Month 1 Day 1
  For participants <5 years of age, palatability will be indirectly assessed by the parent(s)/caregiver(s) of participants using the following: On the basis of the reaction/facial expression of your child, do you think that the medication is (pleasant, not sure, unpleasant)?
Acceptability/Ease of Administration of PTC923 | Month 1 Day 1
  For all participants <12 years of age, parent(s)/caregiver(s) will rate the acceptability/ease of administration, with the following question: Do you sometimes have problems in giving the medication to your child because he/she refuses to take it or throws it up? (Yes/No).
Taste/Flavor Assessment Using a Facial Hedonic Scale | Month 1 Day 1
  For participants ≥5 to <18 years of age who are able to comply with the instructions, the participant will rate the taste/flavor using a facial hedonic scale (5=really good; 4=good; 3=not sure; 2=bad; 1=really bad).
Plasma Sepiapterin Concentration | Month 1 Day 1 up to Month 11 Day 1
Plasma BH4 Concentration | Month 1 Day 1 up to Month 11 Day 1

CONTACTS AND LOCATIONS:
Locations (45):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - UF College of Medicine, Department of Pediatrics Division of Genetics and Metabolism, Gainesville, Florida
  - Indiana University School of Medicine Department of Medical and Molecular Genetics, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai (ISMMS), New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - PARC Clinical Research, Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
- Brazil (2):
  - Hospital de clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
- Canada (3):
  - Metabolics and Genetics in Calgary (MAGIC) Clinic, Ltd., Calgary, Alberta
  - McMaster Children's Hospital Hamilton Health Sciences, Hamilton, Ontario
  - The Hospital for Sick Children University of Toronto Adult Clinic: The Fred A Litwin Family Centre in Genetic Medicine University Health Network & Mt. Sinai Hospital, Toronto, Ontario
- Fakultní nemocnice Královské Vinohrady Klinika dětí a dorostu Ambulance pro léčbu PKU a HPA, Prague, Czechia
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- Hôpital Necker-Enfants Malades - Centre de Référence des Maladies Héréditaires du Métabolisme, Paris, France
- Medical Genetics and Laboratory Diagnostics Center, Tbilisi, Georgia
- Germany (3):
  - University Children's Hospital Hamburg Eppendorf (Kinder-UKE) Klinik für Kinder- und Jugendmedizin (Kinder-UKE), Hamburg
  - Universitätsklinikum Heidelberg / Zentrum für Kinder- und Jugendmedizin / Sektion für Neuropädiatrie & Stoffwechselmedizin, Heidelberg
  - Universitätsklinikum Münster, Münster
- Italy (2):
  - Azienda Ospedaliera-Universita Padova, Padua, Veneto
  - Department of Human Neuroscience, Child and Adolescent Neuropsychiatry, Policlinico Umberto I, Rome
- Japan (3):
  - PTC Clinical Site 1, Multiple Locations
  - PTC Clinical Site 2, Multiple Locations
  - PTC Clinical Site 3, Multiple Locations
- PanAmerican Clinical Research, Guadalajara, Jalisco, Mexico
- UMCG Beatrix Children's Hospital, Groningen, Netherlands
- Pomorski Uniwersytet Medyczny w Szczecinie Centrum Wsparcia Badań Klinicznych, Szczecin, Poland
- Portugal (3):
  - CENTRO HOSPITALAR UNIVERSITÁRIO LISBOA NORTE Hospital de Santa Maria,, Lisbon, Estremadura
  - CENTRO HOSPITALAR UNIVERSITÁRIO LISBOA NORTE Hospital de Santa Maria, Lisbon, Estremadura
  - Centro Hospitalar Universitário Do Porto, Epe, Porto
- Univerzitetni klinicni center Ljubljana, Ljubljana, Slovenia
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona, Esplugues de Llobregat
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Altındağ, Ankara
  - Gazi Üniversitesi Tıp Fakültesi, Yenimahalle, Ankara
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi, Fatih, Istanbul
  - Ege University Faculty of Medicine Children Hospital, Bornova, İzmir
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi, Adana
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - UNIVERSITY HOSPITALS BIRMINGHAM NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital, London